CLINICAL TRIAL: NCT06360380
Title: REFORM-HF™ Reducing Fluid Overload Using Renal Independent SysteM in Heart Failure Patients
Brief Title: Reducing Fluid Overload in Heart Failure Patients Using a Non-invasive, Renal Independent System
Acronym: REFORM-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AquaPass Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AQP-CLP-004
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Heart Failure; CKD Stage 3
Keywords: Aquapass; Sweat Enhancement; Fluid removal; CHF

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, single-arm, within-patient-controlled, pivotal trial, enrolling patients with decompensated heart failure and/or CKD stage 2-3 inadequately responding to current medical treatment, indicated by persistent or worsening congestion despite a daily dose of ≥40 mg furosemide or equivalent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- AquaPass (Experimental): An AquaPass treatment session (up to 5-Hrs.) will be administered in the outpatient settings or at home and supervised by a certified study staff
  Interventions: Device: AquaPass System
- Control (No Intervention): An observation visit, during which data will be collected on fluid intake, fluid output, congestion score, body weight, and quality of life. These data will serve as a control for the efficacy primary endpoint comparison.

INTERVENTIONS:
Device: AquaPass System — a treatment session of up to 5 hours with the AquaPass system, evaluating net fluid removal for efficacy analysis and effect on vital signs for safety analysis
  Arms: AquaPass

SUMMARY:
The REFORM-HF study aims to test a new technology, AquaPass, designed to assist patients experiencing symptoms of fluid overload due to Heart Failure.

Patients will wear a lightweight suit that helps remove excess fluids through their sweat.

The investigators want to see if the AquaPass system can remove an additional 500mL of fluids during treatment, alongside patients' regular medications like diuretics.

Participants will select if to be treated at their home or in the outpatient clinic.

DETAILED DESCRIPTION:
This study is being conducted to demonstrate the safety and effectiveness of the AquaPass System in reducing fluid overload in patients with decompensated heart failure and chronic kidney disease stage 2-3 who are not responding adequately or resistant to current medical treatment.

The study checks if patients' fluid loss as a result of taking diuretics medications is improved when using AquaPass in parallel to this treatment.

The evaluation of success is done by comparing participants' weight before and after the use of the AquaPass system, to evaluate if the system effectively removes excess fluids.

Patients will also have blood and urine tests every morning to check how well their kidneys and heart are functioning.

The first visit will be observation only, without using AquaPass. This will serve as the baseline data. The investigators will compare the data of the AquaPass treatments with this baseline to measure the effectiveness of the system in removing access fluids.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years and < 80 years
* Patient, with known decompensated heart failure and/or CKD stage 2 or more presenting with fluid overload, defined by a congestion score of ≥3, who are not responding adequately or are resistant to current medical treatment as evidenced by persistent or worsening congestion, despite a daily dose of 40 mg furosemide or greater or the equivalent dose of another loop diuretic.
* Patients with no Heart Failure related hospitalization in the past 30 days
* No change in diuretic regimen in the past 7 days
* Baseline NT-proBNP ≥600 pg/mL
* Baseline systolic blood pressure ≥100 mmHg
* Patient is able and willing to provide written informed consent, inclusive of the release of medical information, and Health Insurance Portability and Accountability Act (HIPAA) documentation
* Patient is not participating in any clinical investigation that may interfere with the data collection or the results of this study

Exclusion Criteria:

* Patient considered to be in the acute worsening of heart failure: Requiring ventilation, mechanical support or is clinically unstable requiring pressors, deterioration triggered by arrhythmia, infection, or other medical condition unrelated to fluid overload.
* Patient has any known or visible lower body (non-facial) skin problems (open wounds, ulcers, infections)
* Patient with severe peripheral arterial disease
* Patient is pregnant or planning to become pregnant within the study period, or a lactating woman.
* Renal disease with eGFR <25 ml/min/1.73 m2
* Patients with known hypothalamic disorders
* Patients with known hypohidrosis disorders
* Patients with medical technology dependency (gastric (G) tubes, ventilators etc.)
* Patients with cystic fibrosis
* Patients with active infections
* Inability or unwillingness to comply with the study requirements
* Patients with unstable electrolytes or acid-base balance (per investigator's discretion)
* Known Severe aortic valve or mitral valve stenosis
* History of a heart transplant or actively listed for a heart transplant or LVAD
* Implanted left ventricular assist device or implant anticipated <3 months
* Patients with an active, malignant disease and whose life expectancy is < 6 months (per investigator's discretion)
* Unstable or acutely worsening cardiac or renal conditions (per investigator's discretion)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-01-03 (Estimated); Study Completion 2025-01-29 (Estimated)

PRIMARY OUTCOMES:
AquaPass Performance Evaluation | 5 days
  Average Net Fluid Loss calculated as the difference in weight between pre- and post-AquaPass treatment sessions, in comparison to the Control Day observation.
  Total Average Net Fluid Loss during the Treatment Phase should be ≥ 500gr. as compared to the Total Average Net Fluid Loss during the Control Phase.

SECONDARY OUTCOMES:
AquaPass Safety Evaluation | 6 hours
  Incidence of device-related side effects - defined as events during or up to 1-Hour after device use

CONTACTS AND LOCATIONS:
Overall Officials: Scott C Feitell, DO, Principal Investigator — Rochester Regional Health
Locations (4):
- United States (2):
  - Rochester Regional Health, Rochester, New York
  - Cone Health Advanced Heart Failure Clinic at Moses Cone, Greensboro, North Carolina
- Israel (2):
  - Rambam Medical Campus, Haifa
  - Rabin Medical Center, Petah Tikva